CLINICAL TRIAL: NCT06023342
Title: Examining Engagement Predictors of Health and Fitness App Uptake and Subscription in the General Population: A 24-week Prospective Cohort Study
Brief Title: Examining Engagement Predictors of Health and Fitness App Uptake and Subscription in the General Population
Status: Active, not recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Marc Mitchell, Assistant Professor, Western University, Canada
Other Study IDs: 123207
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Physical Inactivity; Healthy Eating; Mental Health Wellness 1
Keywords: mHealth; behavioural economics; financial incentives; deposit contracts; engagement; physical inactivity; nutrition; mindfullness
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- New users: Approximately 1000 adults (≥18 years old), new to WayBetter app, who have entered into a 7-day free trial, will be studied. Each new user receives a free 1-week trial (that they need to opt into) and $10 USD deposit from WayBetter Inc. They can use the deposit for any game during trial, regardless of continuing membership. To continue to use the app, users pay $69 USD for 6 months. Each game lasts between 1-4 weeks and requires players to achieve a specific behavioural goal. Games require $10-30 deposit, chosen at signup. Validation methods vary; some sync with wearables, others submit activity photos (steps, meals). A user can join up to 10 games simultaneously. "Winners" of each game share deposits, gaining original deposit plus profit, based on 'losses'.

SUMMARY:
This will be a 24-week prospective study that will incorporate user base data of WayBetter Inc.'s app, "WayBetter," to examine user mHealth app engagement. The primary objective of this study is to examine predictors (i.e., socio-demographics, past health behaviours, psychological determinants, app engagement metrics) of (a) initial six-month subscription and b) subscription renewal rates at six months for the WayBetter app. The secondary objective is to characterize WayBetter app engagement over the first 24 weeks of app use.

Participants will be asked to complete a survey that aims to collect the information regarding individual-level socio-demographics, previous health behaviours, and behavioural/personality traits. App engagement metrics will be collected from the WayBetter app.

DETAILED DESCRIPTION:
This will be a 24-week prospective cohort study that will incorporate user base data of WayBetter Inc.'s app, "WayBetter," to examine user mHealth app engagement. Our study sample will consist of approximately 1000 adult users (aged ≥18 years old), who are new app users. As users may have varying registration dates, the data collected will only include the first 24 weeks of an individual's interaction with the platform. To be included, study participants must be enrolled (within five days) and/or recently completed their seven-day free trial on the WayBetter app. Participants who are not proficient in the English language will be excluded. Prior to gaining access to the app, participants must provide informed electronic consent allowing aggregated data (without identifiers) to be shared with third parties, as a part of WayBetter's privacy policy (https://waybetter.com/privacy).

WayBetter is a wellness lifestyle mHealth app available to anyone who wants to improve their overall well-being. All users are asked to accept the company's privacy policy and are prompted to fill out personal data including (but not limited to) [email address, weight] when creating an account. All users are given a one-week free trial as well as $10 USD to use as a deposit towards any WayBetter app game, courtesy of WayBetter Inc. Users can complete any of the games they signed up for during their free trial, even if they decide not to continue to their membership. To continue to participate in games, users must subscribe to a six-month membership ($69 USD total). In general, users can join up to ten games at a time. The app has a game directory ("explore" tab) that includes 60+ games each week in three categories: fitness, nutrition, and mindset. New games start on Mondays, Wednesdays, and Fridays. Each game lasts between 1-4 weeks and requires players to achieve a specific behavioral goal (e.g., 5K Steps Per Day requires that they walk at least 5,000 steps per day on at least four days per week for two weeks). Another example of a game would be, "Healthy Hacks" which requires participants to focus on portion control and finding healthier alternatives to snacks on at least two days during the week. Or "Read A Book" which encourages participants to unwind with a 15-minute reading session on at least four days per week for two weeks. Upon joining a game, players have an option to make a deposit, called a "financial commitment" of $10-30, depending on the game. Multiple methods are used to validate goal achievement. Some games require players to verify their physical activity data by connecting their WayBetter app account (i.e., syncing) to a wearable device or step tracking app. Other games require participants to verify their behavior by submitting photos (e.g., photo from their wearable device or step tracking app showing that they met the game's daily step goal; photo of meals they ate). Each game also has a social feed, where users can view each other's posts and photo submissions and share anything related to their fitness journey (e.g., progress, inspiration, something they are proud of). All players who achieve the game's goal are declared "winners." Winners who made deposits are rewarded by splitting the total pot of deposits evenly, such that they earn back their original deposit plus addition profit, dependent on how many users 'lost'. The app incorporates an additional gamification aspect by introducing levels; players are required to win 3 games to advance a level (one from each category; they can choose any games they want).

WayBetter will send out a recruitment email to WayBetter users five days after they enter into a seven-day free trial. A reminder email will be sent to users seven day after the initial recruitment email was sent (day 12 of account creation) to prompt survey completion. A free trial sign-up for the WayBetter app can occur in two ways. First, a user completing the WayBetter "quiz" (a survey marketed via social media platforms and on the WayBetter website; Group A, "quiz taker"), can sign up at the end of the survey to begin their 'personalized journey' to healthy living (based on their survey answers) by starting their free seven-day trial. The user would then place their credit card information to secure their 'personalized journey', create an account, and begin their seven-day free trial. The second method to begin a free trial is when a user has already downloaded the app (Group B, "organic" users), created an account, and then is prompted by the app to provide their credit card information to sign up for a seven-day free trial. In this recruitment email, participants will be invited to complete a study survey via the RedCAP link provided. Participants will be prompted to complete the survey within five days to create urgency to complete the quiz. We want new users to complete the survey as soon as possible from the time they completed the free trial, so that they do not become an experienced user, which has the potential to affect the way they answer some of the survey questions. After clicking on the link, participants will first be prompted to read the study LOI. Thereafter, participants will be asked to complete the survey which will aim to collect information about individual-level socio-demographics (i.e., household income, rural or urban living status, gender, age, race, and ethnicity), previous health behaviours (i.e., previous fitness, nutrition, stress, weight loss), determinants of behavioural intentions to use health and fitness apps, and behavioural/personality traits (i.e., risk taking traits, healthy behaviour self-efficacy, personality traits). Participants who complete the survey will earn a $10 USD Amazon e-gift card, distributed to their participant provided email within ten days of completion.

Any games that did not utilize deposit wagers (i.e., accountability partners or no motivational booster) will not be included in the analysis. Our primary outcomes are rates of (a) initial six-month subscription and b) subscription renewal rates at six months, for the WayBetter app. User' specific metrics, 'psychological' metrics, and app engagement ('WayBetter' and 'Industry' specific) metrics of users who sign up for the 6-month subscription will be used to identify underlying homogenous subgroups of individuals using Latent Class Analysis (LCA). Next, associations between the subgroups (termed 'latent classes') to determine which users are more likely to sign-up, subscribe, and renew subscription to the WayBetter app will be examined. Linear regressions and Cox Proportional Hazard regression models to examine engagement correlates will be used. Post Hoc analysis will be used to determine between which users the statistical differences lie. The secondary objective is to describe WayBetter app engagement over 24 weeks using 'WayBetter' and 'Industry' specific engagement metrics. Descriptive statistics to summarize engagement patterns and Kaplan-Meier survival curves to illustrate time to non-usage attrition and app resumption will be used. A repeated measures ANOVA will be used to demonstrate if statistically significant differences exist between the user 'latent classes' and app engagement metrics. Regression equations and a linear probability model will be formed to predict engagement metrics using latent classes and individual-level factors (sociodemographic, previous health behaviours, determinants of behavioural intentions to use health and fitness apps, and behavioural/personality traits) as predictor variables. A sensitivity analysis will be completed to examine the effects of methods of WayBetter account creation, 1) via the WayBetter online quiz (Group A) or 2) direct download of the app on primary outcomes (Group B).

ELIGIBILITY:
Inclusion Criteria:

* WayBetter Inc.'s users who enrolled and/or recently completed (within five days) their seven-day free trial on the WayBetter app
* User's are must be 18 years or older.

Exclusion Criteria:

* Users under the age of 18 are excluded to ensure that the sample represents to an adult demographic
* Users who are unable to communicate in English are excluded as the survey necessitates completion in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study cohort comprises individuals who register an account on the WayBetter app and successfully finish the survey within the recruitment timeframe.
Sampling Method: Non-Probability Sample
Enrollment: 1084 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Six-month Subscription | Day one of seven-day free trial [Week One] to end of seven-day free trial [End of Week One]
  Total number of six-month WayBetter subscriptions started after a free trial
Subscription Renewal Rates | Week 24
  Measured by number of subscription renewal rates after 6 months

SECONDARY OUTCOMES:
App opens per week | Week 1 to Week 24
  Number of app opens for one second or longer
Date of Joining First Game | Measured between Week 1 to Week 24
  Number of days from joining free trial to joining first game
Game Adherence | Week 1 to Week 24
  Number of verifications submitted during a game vs number of verifications required by WayBetter game
Number of games started and won each week | Week 1 to Week 24
  Total number of games by (a) category (b) type (c) verification method and (d) earnings started and won each week
Non-usage attrition | First occurrence of four weeks of inactivity
  Number of no app opens [one second or longer] for four weeks or longer
Re-engagement | First occurrence of two consecutive weeks of app opens
  First occurrence of two weeks of app resumption [one app one of one second or longer for two consecutive week]

CONTACTS AND LOCATIONS:
Overall Officials: Marc Mitchell, PhD, Principal Investigator — Western University
Locations (1):
- University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No